CLINICAL TRIAL: NCT03940534
Title: Utilization of the TAD Device for Dispensing Pain Medications in Hospice Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intent Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 6195-001
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Medication Adherence; Satisfaction, Personal
MeSH Terms: conditions — Medication Adherence; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This study is a randomized crossover design.
Masking Description: No masking is to be used in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Start with Mobile Device (Active Comparator)
  Interventions: Device: TAD
- Start without Mobile Device (Active Comparator)
  Interventions: Device: TAD

INTERVENTIONS:
Device: TAD — TAD is a device used to aid medication adherence.

SUMMARY:
A novel device, TAD, has been developed to aid adherence to prescribed regimens and may have a roll in hospice pain management. This study aims to assess medication adherence relating to missed doses or improperly timed doses with and without the aid of a mobile device as a primary endpoint. Secondary endpoints will be patient, nursing, and provider satisfaction.

DETAILED DESCRIPTION:
This study is a randomized crossover study in which patients will be randomized to start with or without a mobile device assisting the patient or caregiver in using the device. The investigators aim to enroll 20 patients across 3 sites. Each patient is expected to participate in the study for 12 weeks. After the first 2 weeks of participation, the patient will either begin using the mobile device to assist or will stop using the mobile device for the next 2 weeks. after the initial 4 weeks, the patient will choose to continue with or without using the mobile device.

ELIGIBILITY:
Inclusion Criteria:

* any patient taking morphine ER or Oxycontin on one of three hospice home teams

Exclusion Criteria:

* pregnancy
* inability to demonstrate competent use of the device
* age less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Difference from Scheduled Dosing Time | through study completion, up to 1 year
  The time difference between when the patient took the dose and the scheduled time of administration.
Missed Doses | through study completion, up to 1 year
  The number of missed doses that occurred during the study.

SECONDARY OUTCOMES:
Patient Satisfaction: scale of 1 to 5 | through study completion, up to 1 year
  The patient's satisfaction will be measured on a scale of 1 to 5 (from 1 being extremely dissatisfied to 5 being extremely satisfied). Satisfaction will be assessed with the follow questions:
  1. Using the mail order pharmacy to receive your pain medication?
  2. Ease of using the TAD device to dispense your pain medication?
  3. Ease of using the mobile device application with the TAD device? (ONLY when using the mobile application)
  4. The ability of the device to provide you the dose of pain medication at the correct time?
  5. The overall experience of using the TAD device?
Nurse Satisfaction: scale of 1 to 5 | through study completion, up to 1 year
  The nurse's satisfaction will be measured on a scale of 1 to 5 (from 1 being extremely dissatisfied to 5 being extremely satisfied). Satisfaction will be assessed with the follow questions:
  1. Using the mail order pharmacy get your patient their pain medication?
  2. Your patient's ability to use the TAD device to dispense their pain medication?
  3. Your patient's ability to use the mobile device application with the TAD device? (ONLY when using the mobile application)
  4. The ability of the device to increase compliance of the pain medication?
  5. The overall experience of using the TAD device?
Physician Satisfaction: scale of 1 to 5 | through study completion, up to 1 year
  The physician's satisfaction will be measured on a scale of 1 to 5 (from 1 being extremely dissatisfied to 5 being extremely satisfied). Satisfaction will be assessed with the follow questions:
  1. Using the mail order pharmacy get your patient their pain medication?
  2. Your patient's ability to use the TAD device to dispense their pain medication?
  3. Your patient's ability to use the mobile device application with the TAD device? (ONLY when using the mobile application)
  4. The ability of the device to increase compliance of the pain medication?
  5. The overall experience of using the TAD device?satisfaction will be measured on a scale of 1 to 5 for satisfaction of using the mail order pharmacy, ease of using the device, ease of using the mobile device, the ability of the device to accurately provide the dose, and overall experience with the device.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Richter, PharmD, Principal Investigator — Clinical Pharmacist; Ellen Talos, MD, Study Director — Medical Director
Locations (3):
- United States (3):
  - Haven: Advanced Illness Care, Gainesville, Florida
  - Haven: Advanced Illness Care, Lake City, Florida
  - Haven: Advanced Illness Care, Palatka, Florida

IPD SHARING:
Plan to Share IPD: Undecided
Other study staff may apply to access the data through an appropriate IRB in the future, but this is not known at this time.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03940534/Prot_SAP_000.pdf